CLINICAL TRIAL: NCT04707469
Title: Efficacy and Safety of Once-daily Oral Semaglutide 25 mg and 50 mg Compared With 14 mg in Subjects With Type 2 Diabetes
Brief Title: Research Study to Compare Three Doses of Semaglutide Tablets Taken Once Daily in People With Type 2 Diabetes
Acronym: PIONEER PLUS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9924-4635; U1111-1247-0210 (Other: World Health Organization (WHO)); 2020-000299-39 (Registry Identifier: European Medicines Agency (EudraCT))
Record Dates: First submitted 2021-01-12; First posted 2021-01-13 (Actual); Results first posted 2024-04-03 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Oral semaglutide 50 mg (Experimental): Participants will receive once daily semaglutide tablets in a dose escalating manner for 68 weeks: 3 mg (week 1-4), 7 mg (week 5-8), 14 mg (week 9-12), 25 mg (week 13-16) and 50 mg (week 17-68).
  Interventions: Drug: Oral semaglutide
- Oral semaglutide 25 mg (Experimental): Participants will receive once daily semaglutide tablets in a dose escalating manner for 68 weeks: 3 mg (week 1-4), 7 mg (week 5-8), 14 mg (week 9-12) and 25 mg (week 13-68).
  Interventions: Drug: Oral semaglutide
- Oral semaglutide 14 mg (Active Comparator): Participants will receive once daily semaglutide tablets in a dose escalating manner for 68 weeks: 3 mg (week 1-4), 7 mg (week 5-8) and 14 mg (week 9-68).
  Interventions: Drug: Oral semaglutide

INTERVENTIONS:
Drug: Oral semaglutide — Participants will receive once daily semaglutide tablets (oral administration) in a dose escalating manner for 68 weeks.

SUMMARY:
This study compares three doses of once daily semaglutide tablets in people with type 2 diabetes who were previously treated with other oral anti-diabetic medicines. Participants will be initiated on the lowest starting dose of 3 mg and gradually increased until they reach the final trial dose of 14 mg, 25 mg or 50 mg once daily semaglutide tablets. The final three doses will be randomized (i.e., decided by chance). Participants will be administered one tablet per day for 68 weeks. Women cannot take part if they are pregnant, breast-feeding or planning to become pregnant during the study period. Women who can get pregnant will be checked for pregnancy via urine tests. Once daily semaglutide tablets (3 mg, 7 mg and 14 mg) are approved for the treatment of type 2 diabetes in the US, in the EU and in some other countries, under the brand name Rybelsus®.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age above or equal to 18 years at the time of signing informed consent.
* Diagnosed with type 2 diabetes mellitus at least 180 days prior to the day of screening.
* HbA1c of 8.0-10.5% (64-91 mmol/mol) (both inclusive).
* BMI equal to or above 25 kg/m^2
* Stable daily dose(s) for 90 days prior to the day of screening of any of the following treatment regimens:
* No more than 3 of the following oral anti-diabetic drugs and at least 1 marked with a *:

  * Metformin (equal to or above1500 mg or maximum tolerated or effective dose).
  * Sulfonylureas (SU) (equal to or above half of the maximum approved dose according to local label or maximum tolerated or effective dose).
  * Sodium/glucose cotransporter 2 (SGLT2) inhibitors (maximum tolerated dose).
* Dipeptidyl peptidase-4 (DPP-4) inhibitors (maximally indicated dose as per local label).
* Subjects, on treatment with stable dose of DPP-4 inhibitors at inclusion, must be willing to discontinue DPP-4 inhibitor treatment at randomisation (with no wash-out).

Exclusion Criteria:

* Treatment with any medication indicated for the treatment of diabetes or obesity other than stated in the inclusion criteria within the past 90 days prior to the day of screening. However, short term insulin treatment for a maximum of 14 days prior to the day of screening is allowed.
* Renal impairment measured as estimated glomerular filtration rate (eGFR) value of below 30 mL/min/1.73 m^2 according to Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) creatinine equation as defined by kidney disease improving global outcomes (KDIGO 2012) classification.
* Uncontrolled and potentially unstable diabetic retinopathy or maculopathy. Verified by a fundus examination performed within the past 90 days prior to screening or in the period between screening and randomisation. Pharmacological pupil-dilation is a requirement unless using a digital fundus photography camera specified for non-dilated examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1606 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2023-03-07 (Actual); Study Completion 2023-03-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 1452), Study Director — Novo Nordisk A/S
Locations (226):
- United States (82):
  - American Clinical Trials, Buena Park, California
  - Valley Research, Fresno, California
  - Velocity Clin Res San Diego, La Mesa, California
  - First Valley Medical Group, Lancaster, California
  - Pacific Clinical Studies, Los Alamitos, California
  - Velocity Clin Res Los Angeles, Los Angeles, California
  - Diabetes Medical Center Of California, Northridge, California
  - Desert Oasis Hlthcr Med Group, Palm Springs, California
  - Gateway Research Center, Poway, California
  - Encompass Clinical Research_Spring Valley, Spring Valley, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - San Fernando Valley Hlth Inst, LLC, West Hills, California
  - University of Colorado Hospital, Aurora, Colorado
  - Optumcare Clinical Trials,LLC-Golden, Colorado Springs, Colorado
  - Chase Medical Research LLC, Waterbury, Connecticut
  - Alliance for Multispec Res, Coral Gables, Florida
  - Northeast Research Institute, Jacksonville, Florida
  - San Marcus Res Clin Miami Lakes, Miami Lakes, Florida
  - Complete Health Research, Ormond Beach, Florida
  - Clinical Trial Res Assoc,Inc, Plantation, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Endo Res Solutions Inc, Roswell, Georgia
  - East West Med Res Inst, Honolulu, Hawaii
  - Elite Clinical Trials, Blackfoot, Idaho
  - Rocky Mt Clin Res, LLC, Idaho Falls, Idaho
  - Solaris Clinical Research, Meridian, Idaho
  - Cedar-Crosse Research Center, Chicago, Illinois
  - Macoupin Research Group, Gillespie, Illinois
  - UnityPoint Health-Diabetes Care Center, Peoria, Illinois
  - Evanston Premier Hlthcr Res, Skokie, Illinois
  - Midwest Inst For Clin Res, Indianapolis, Indiana
  - Iowa Diab & Endo Res Center, West Des Moines, Iowa
  - Cotton O'Neil Diab & Endo Ctr, Topeka, Kansas
  - The Research Group of Lexington LLC, Lexington, Kentucky
  - L-MARC Research Center, Louisville, Kentucky
  - Pennington Biom Res Ctr, Baton Rouge, Louisiana
  - Centex Studies, Inc._Lake Charles, Lake Charles, Louisiana
  - MD Medical Research, Oxon Hill, Maryland
  - Brigham & Women's Hospital, Boston, Massachusetts
  - MassResearch, LLC, Waltham, Massachusetts
  - Aa Mrc Llc, Flint, Michigan
  - Arcturus Healthcare, PLC., Troy, Michigan
  - Mercury Str Med Grp, PLLC, Butte, Montana
  - Univ of Nebraska Medical CTR, Omaha, Nebraska
  - University of Nebraska Medical Center-Diabetes Center, Omaha, Nebraska
  - Premier Research Inc., Trenton, New Jersey
  - UNC Diabetes Care Center_Chapel Hill, Chapel Hill, North Carolina
  - PharmQuest Life Sciences LLC, Greensboro, North Carolina
  - Accellacare, Wilmington, North Carolina
  - Lillestol Research LLC, Fargo, North Dakota
  - Rapid Medical Research Inc, Cleveland, Ohio
  - Prestige Clinical Research, Franklin, Ohio
  - Albert J Weisbrot, Mason, Ohio
  - Intend Research, Norman, Oklahoma
  - Corvallis Clinic PC Clinical Research Department, Corvallis, Oregon
  - Preferred Primary Care Physicians_Pittsburgh, Pittsburgh, Pennsylvania
  - Palmetto Clinical Research, Greenville, South Carolina
  - Palmetto Clinical Research, Summerville, South Carolina
  - Holston Medical Group Pc, Bristol, Tennessee
  - Chattanooga Medical Research, LLC, Chattanooga, Tennessee
  - Murphy Research Center, Humboldt, Tennessee
  - Clinical Neuroscience Solutions, Memphis, Tennessee
  - Arlington Family Res. Ctr Inc, Arlington, Texas
  - Velocity Clinical Res-Dallas, Dallas, Texas
  - Velocity Clinical Research, Dallas, Dallas, Texas
  - UT Southwestern Med Cntr, Dallas, Texas
  - Care United Research, LLC, Forney, Texas
  - JCCT- Juno NW Houston, Houston, Texas
  - Southwest Clinical Trials, Houston, Texas
  - Family Practice Care Associates, Humble, Texas
  - Research Trials Worldwide LLC, Humble, Texas
  - Juno Research, LLC_Cary, Katy, Texas
  - DCOL Ctr for Clin Res, Longview, Texas
  - Research Institute Of Dallas, Plano, Texas
  - VIP Trials, San Antonio, Texas
  - Consano Clinical Research, LLC, Shavano Park, Texas
  - Simcare Medical Research, LLC, Sugar Land, Texas
  - Health Res of Hampton Roads, Newport News, Virginia
  - York Clinical Research LLC, Norfolk, Virginia
  - Dominion Medical Associates, Richmond, Virginia
  - Capital Clin Res Ctr,LLC, Olympia, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
- Australia (7):
  - Liverpool Hospital, Liverpool, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Core Research Centre, Milton, Queensland
  - South Australian Endocrine Research, Keswick, South Australia
  - Southern Adelaide Diabetes & Endocrine Services, Oaklands Park, South Australia
  - Barwon Health (The Geelong Hospital), Geelong, Victoria
  - Fremantle Hospital, Fremantle, Western Australia
- Bulgaria (17):
  - MHAT - Blagoevgrad AD, Department of Internal Diseases, Blagoevgrad
  - Medical Center Zdrave Lom EOOD, Lom
  - UMHAT Pulmed OOD - Pazardzhik, Department of Internal Diseases, Pazardzhik
  - "MHAT - Pazardzhik", Pazardzhik
  - OCSOMCE - Dr. Albena Dinkova EOOD, Pleven
  - UMHAT Kaspela EOOD, Endocrinology and Metabolic Diseases Clinic, Plovdiv
  - MHAT Sveta Karidad EAD, Plovdiv
  - MHAT Hadzhi Dimitar OOD, Sliven
  - Medical center Smolyan clinical research OOD, Smolyan
  - UMHAT "Aleksandrovska", Sofia
  - USHATE "Akad. Ivan Penchev" Second Clinic of Endocrinology, Sofia
  - Medical Institute of Ministry of interior, Sofia
  - UMHAT Sveta Marina EAD, Varna
  - AIPSMC Dr. Artin Magardichyan EOOD, Varna
  - MHAT- Hristo Botev AD, Vratsa
  - MHAT- Hristo Botev, Vratsa
  - MHAT Sveti Panteleimon - Yambol AD, Yambol
- Canada (15):
  - LMC Clin Res Inc. Calgary, Calgary, Alberta
  - C-endo Diab Endo Clin Calgery, Calgary, Alberta
  - G.A. Research Associates Ltd., Moncton, New Brunswick
  - LMC ClinRsrh Inc.Brampton, Brampton, Ontario
  - LMC Clinical Res Thornhill, Concord, Ontario
  - LMC Endo Ctr (Etobicoke) Ltd, Etobicoke, Ontario
  - Wharton Med Clin Trials, Hamilton, Ontario
  - LMC Research Inc. Ottawa, Nepean, Ontario
  - LMC Oakville, Oakville, Ontario
  - Stayner Medical Clinic, Stayner, Ontario
  - Winterberry Family Medicine, Stoney Creek, Ontario
  - LMC Endo Centres Ltd.(Bayview), Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Applied Med Inf Res, Montreal, Quebec
  - LMC Clin Rsrch Inc. (Montreal), Saint-Laurent, Quebec
- Croatia (7):
  - Poliklinika Solmed, Zagreb, City of Zagreb
  - KBC Rijeka, Endokrinologija, Rijeka, Primorje-Gorski Kotar County
  - Opca bolnica Bjelovar, Bjelovar
  - Klinicki bolnicki centar Osijek, Osijek
  - General Hospital Dr. Josip Bencevic_Diabetic department, Slavonski Brod
  - KB Dubrava, Zavod za endokrinologiju i dijabetes, Zagreb
  - Klinicka bolnica Sveti Duh, Zagreb
- Czechia (9):
  - Ordinace pro choroby srdce, Chomutov
  - Diabetologická a endokrinologická ambulance Hlučín, Hlučín
  - Diahaza s.r.o., Holešov
  - Diahelp - diabetologie, Pardubice
  - DIALINE s.r.o., Plzeň 3
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - DiaGolfova spol s.r.o., Prague
  - Diabet2 s.r.o., Prague
  - Diabetologická a endokrinologická ambulance Praha, Prague
- Estonia (6):
  - Private Endocrnologist Dr Viitas, Pärnu
  - East Tallinn Central Hospital, Tallinn
  - Merelahe Family Doctors Centre, Tallinn
  - Estonian Diabetes Centre, Tallinn
  - Tartu University Hospital Internal Medicine Clinic, Tartu
  - SA Viljandi Haigla, Viljandi
- Germany (8):
  - Institut für Klinische Forschung und Entwicklung, Berlin
  - Plassmann, Essen
  - Zentrum für klinische Forschung, Dr. med. Lüdemann, Falkensee
  - Diabetes Zentrum Wandsbek Berufsausuebungsgemeinschaft GbR, Hamburg
  - Wendisch/Dahl Hamburg (DZHW), Hamburg
  - Institut für Diabetesforschung GmbH Münster - Dr. med. Rose, Münster
  - RED-Institut für medizinische Forschung und Fortbildung GmbH, Oldenburg in Holstein
  - Praxis Dr. med. Wenzl-Bauer, Rehlingen-Siersburg
- Hungary (11):
  - PTE-AOK II. Belgyogyaszati Klinika es Nephrologiai Centrum, Pécs, Baranya Vármegye
  - Komáromi Selye János Kórház, Komárom, Komárom-Esztergom
  - Óbudai Egészségügyi Centrum, Budapest, Pest County
  - Szőcs Depot Egészségügyi Szolgáltató Kft., Budapest
  - Bajcsy-Zsilinszky Kórház, Budapest
  - Dr. Vass László Egészségügyi Intézmény Diab. Szakrendelés, Budapest
  - Debreceni Egyetem Klinikai Központ Belgyógyászati Klinika D épület, Debrecen
  - Debreceni Egyetem Klinikai Központ Belgyógyászati Klinika, Debrecen
  - Tolna megyei Balassa János Kórház, Szekszárd
  - Fejér Megyei Szent György Oktatókórház, Székesfehérvár
  - Vas Vármegyei Markusovszky Egyetemi Oktatókórház, Szombathely
- India (25):
  - Endolife Specialty Hospitals, Guntur, Andhra Pradesh
  - Care Outpatient Centre, Hyderabad, Andhra Pradesh
  - Kurnool Medical Collage, Kurnool, Andhra Pradesh
  - Nirmal Hospital Pvt. Ltd., Surat, Gujarat
  - PGIMS Rohtak, Rohtak, Haryana
  - Ramaiah Memorial Hospital, Bangalore, Karnataka
  - Belgaum Diabetes Centre, Belagavi, Karnataka
  - KLES & Prabhakar Kore Hospital and Research Centre, Belagavi, Karnatka
  - Amrita Institute Of Medical Sciences & Research Centre, Kochi, Kerala
  - Seth GS medical college and KEM Hospital, Mumbai, Maharashtra
  - Apollo Hospital, Navi Mumbai, Mumbai, Maharashtra
  - Deenanath Mangeshkar Hospital & Research Centre, Pune, Maharashtra
  - Deenanath Mangeshkar Hospital and Research Centre, Pune, Maharashtra
  - Inamdar Multispeciality Hospital, Pune, Maharashtra
  - Fortis Hospital, Shalimar Bagh, New Delhi, New Delhi, National Capital Territory of Delhi
  - Apollo Hospital, Delhi, New Delhi
  - All India Institute of Medical Sciences, New Dehli, New Delhi
  - Dayanand Medical College & Hospital, Ludhiana, Punjab
  - Christian Medical College Hospital, Vellore, Vellore, Tamil Nadu
  - Gandhi Hospital & Medical college, Hyderabad, Telangana
  - Gleneagles Hospitals, Hyderabad, Telangana
  - Osmania General Hospital, Hyderabad, Telangana
  - MV Hospital and Research Centre, Lucknow, Uttar Pradesh
  - I.P.G.M.E & R Hospital, Kolkata, West Bengal
  - Apollo Multispeciality Hospital, Kolkata, Kolkata, West Bengal
- Poland (21):
  - NZOZ Przychodnia Specjalistyczna Medica, Lublin, Lubelski
  - Specjalistyczny Gabinet Diabetologiczny Radoslaw Rumianowski, Gorzów Wielkopolski, Lubusz Voivodeship
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Bialystok, Podlaskie Voivodeship
  - NZOZ Specjalistyczny Osrodek Internistyczno-Diabetologiczny Małgorzata Arciszewska, Bialystok, Podlaskie Voivodeship
  - Kresmed Sp. z o. o., Bialystok, Podlaskie Voivodeship
  - Centrum Zdrowia Metabolicznego, Poznan, Wielkopolskie Voivodeship
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Bialystok
  - Osteo Medic s.c. Artur Racewicz Jerzy Supronik, Bialystok
  - SNZOZ Lege Artis, Bialystok
  - Centrum Kliniczno Badawcze, Elblag
  - Centrum Badan Klinicznych PI-House, Gdansk
  - Uniwersyteckie Centrum Kliniczne im. prof. Gibinskiego, SUM, Katowice
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Szpital Uniwersytecki w Krakowie, Krakow
  - Centrum Terapii Wspolczesnej J.M. Jasnorzewska S.K.A., Lodz
  - Gaja Poradnie Lekarskie, Poznan
  - Centrum Medyczne "Diabetika", Radom
  - NBR Polska Tomasz Klodawski, Warsaw
  - SP CSK Klinika Diabetologii i Chorob Wewnetrznych, Warsaw
  - Panstwowy Instytut Medyczny Ministerstwa Spraw Wewnetrznych I Administracji, Warsaw
  - Centrum Medyczne Oporow, Wroclaw
  - Prywatny Gabinet Janusz Gumprecht, Zabrze
- Manati Ctr For Clin Research, Manatí, Puerto Rico
- Slovakia (10):
  - DIADA, s.r.o., Bardejov
  - Diabetologicka ambulancia Diabetes care, s.r.o., Hnúšťa
  - Diabetologicka ambulancia DIAMO s.r.o., Kežmarok
  - MOMED, s.r.o, Kráľovský Chlmec
  - IN-DIA s.r.o., Lučenec
  - Diabetologicka ambulancia MUDr. Alena Lomencikova, s.r.o, Martin
  - DIABETOL, s.r.o., Prešov
  - OLIVER - MED s.r.o., Rimavská Sobota
  - MEDI-DIA s.r.o., Sabinov
  - Diabetologicka ambulancia MUDr. Gabriela Zimova, Spišská Nová Ves
- Slovenia (5):
  - General Hospital Celje, Celje
  - Healthcare Centre Koper, Koper
  - UKC Ljubljana, Endocrinology and Diabetes, Ljubljana
  - UKC Maribor - diabetes, Maribor
  - Healthcare Centre Nova Gorica, Nova Gorica
- Taiwan (2):
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Result] Aroda VR, Aberle J, Bardtrum L, Christiansen E, Knop FK, Gabery S, Pedersen SD, Buse JB. Efficacy and safety of once-daily oral semaglutide 25 mg and 50 mg compared with 14 mg in adults with type 2 diabetes (PIONEER PLUS): a multicentre, randomised, phase 3b trial. Lancet. 2023 Aug 26;402(10403):693-704. doi: 10.1016/S0140-6736(23)01127-3. Epub 2023 Jun 26. PMID 37385279

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted in 14 countries (184 sites screened/177 randomised participants) as follows: Australia: 7/6; Bulgaria: 15/15; Canada: 13/13; Croatia: 5/5; Czech Republic: 5/5; Estonia: 6/5; Germany: 8/8; Hungary: 9/9; India: 20/20; Poland: 18/18; Slovakia: 9/9; Slovenia: 5/5; Taiwan: 2/2; United States: 62/57. In addition, Bulgaria (1 site), Canada (1 site), Croatia (1 site) and Poland (1 site) were approved by the institutional review board, but did not randomise any participant.
Pre-assignment Details: Participants were randomized in 1:1:1 ratio to receive either 14 milligram (mg), 25 mg or 50 mg oral semaglutide once daily. The trial had a 68-week treatment period (8-16 weeks of dose escalation period and 52-60 weeks of maintenance period), followed by a 5-week follow-up period.
Groups:
- Oral Semaglutide 14 mg: Participants were to take oral semaglutide tablets once daily in a dose escalation manner from week 0 to week 68: 3 mg from week 0 to week 4, 7 mg from week 4 to week 8 and 14 mg from week 8 to week 68.
- Oral Semaglutide 25 mg: Participants were to take oral semaglutide tablets once daily in a dose escalation manner from week 0 to week 68: 3 mg from week 0 to week 4, 7 mg from week 4 to week 8, 14 mg from week 8 to 12 and 25 mg from week 12 to week 68.
- Oral Semaglutide 50 mg: Participants were to take oral semaglutide tablets once daily in a dose escalation manner from week 0 to week 68: 3 mg from week 0 to week 4, 7 mg from week 4 to week 8, 14 mg from week 8 to 12, 25 mg from week 12 to week 16 and 50 mg from week 16 to week 68.
Period: Overall Study
Arm/Group | Oral Semaglutide 14 mg | Oral Semaglutide 25 mg | Oral Semaglutide 50 mg
Started | 536 | 535 | 535
Treated | 534 | 534 | 534
Full Analysis Set (FAS) | 536 | 535 | 535
Safety Analysis Set (SAS) | 534 | 534 | 534
Completed | 507 | 490 | 505
Not Completed | 29 | 45 | 30
Not completed — Site closure | 0 | 2 | 0
Not completed — Physician Decision | 2 | 2 | 2
Not completed — Death | 1 | 6 | 2
Not completed — Lost to Follow-up | 9 | 19 | 14
Not completed — Withdrawal by Subject | 17 | 16 | 12

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomised participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Semaglutide 14 mg | Oral Semaglutide 25 mg | Oral Semaglutide 50 mg | Total
Number analyzed (Participants) | 536 | 535 | 535 | 1606
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.4 (10.4) | 58.8 (10.7) | 57.6 (11.2) | 58.2 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 211 | 231 | 228 | 670
  Male | 325 | 304 | 307 | 936
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 38 | 37 | 36 | 111
  Not Hispanic or Latino | 498 | 498 | 499 | 1495
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 85 | 73 | 111 | 269
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 0 | 2
  Black or African American | 19 | 22 | 18 | 59
  White | 424 | 432 | 398 | 1254
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 7 | 6 | 8 | 21

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycated Haemoglobin (HbA1c) (Week 52)
Description: Change from baseline (week 0) in glycosylated haemoglobin (HbA1c) was evaluated at week 52. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of additional anti-diabetic medication or discontinuation of trial treatment. Percentage point refers to arithmetic difference between two percentages.
Time Frame: Baseline (week 0), week 52
Population: Full Analysis Set (FAS) which comprised all randomised participants. Overall number of participants analyzed = participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percentage point of HbA1c
Arm/Group | Oral Semaglutide 14 mg | Oral Semaglutide 25 mg | Oral Semaglutide 50 mg
Number analyzed (Participants) | 497 | 475 | 492
Percentage point of HbA1c | -1.5 (1.3) | -1.9 (1.3) | -2.1 (1.4)
Statistical Analysis 1: Comparison: Oral Semaglutide 14 mg vs Oral Semaglutide 25 mg; Treatment policy estimand; Test type: Superiority — Change from baseline was analyzed using an ANCOVA model with treatment, strata and region as categorical fixed effects and baseline value as covariate for each of the 1000 imputed complete datasets,and pooled by Rubin's rule to draw inference; p = 0.0006, ANCOVA — Unadjusted two-sided p-value for test of no difference; Treatment difference = -0.27, 95% CI 2-sided [-0.42 to -0.12]
Statistical Analysis 2: Comparison: Oral Semaglutide 14 mg vs Oral Semaglutide 50 mg; Treatment policy estimand; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < .0001, ANCOVA — Unadjusted two-sided p-value for test of no difference; Treatment difference = -0.53, 95% CI 2-sided [-0.68 to -0.38]

2. Secondary Outcome: Change From Baseline in Body Weight (Week 52)
Description: Change from baseline (week 0) in body weight was evaluated at week 52. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of additional anti-diabetic medication or discontinuation of trial treatment.
Time Frame: Baseline (week 0), week 52
Population: FAS which comprised all randomised participants. Overall number of participants analyzed = participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: Kilogram (Kg)
Arm/Group | Oral Semaglutide 14 mg | Oral Semaglutide 25 mg | Oral Semaglutide 50 mg
Number analyzed (Participants) | 503 | 480 | 495
Kilogram (Kg) | -4.4 (5.2) | -7.1 (6.8) | -8.3 (7.5)

3. Secondary Outcome: Change From Baseline in HbA1c (Week 68)
Description: Change from baseline (week 0) in HbA1c was evaluated at week 68. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of additional anti-diabetic medication or discontinuation of trial treatment. Percentage point refers to arithmetic difference between two percentages.
Time Frame: Baseline (week 0), week 68
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage point of HbA1c
Arm/Group | Oral Semaglutide 14 mg | Oral Semaglutide 25 mg | Oral Semaglutide 50 mg
Number analyzed (Participants) | 487 | 469 | 491
Percentage point of HbA1c | -1.5 (1.3) | -1.8 (1.3) | -2.0 (1.4)

4. Secondary Outcome: Change From Week 12 in HbA1c (Week 52)
Description: Change in HbA1c was evaluated from week 12 to week 52. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of additional anti-diabetic medication or discontinuation of trial treatment. Percentage point refers to arithmetic difference between two percentages.
Time Frame: Week 12, Week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage point of HbA1c
Arm/Group | Oral Semaglutide 14 mg | Oral Semaglutide 25 mg | Oral Semaglutide 50 mg
Number analyzed (Participants) | 333 | 345 | 339
Percentage point of HbA1c | -0.4 (1.2) | -0.8 (1.1) | -1.0 (1.2)

5. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) (Week 52)
Description: Change from baseline (week 0) in fasting plasma glucose (FPG) was evaluated at week 52. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of additional anti-diabetic medication or discontinuation of trial treatment.
Time Frame: Baseline (week 0), week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: millimole per litre (mmol/L)
Arm/Group | Oral Semaglutide 14 mg | Oral Semaglutide 25 mg | Oral Semaglutide 50 mg
Number analyzed (Participants) | 494 | 460 | 482
millimole per litre (mmol/L) | -2.4 (3.4) | -3.0 (3.5) | -3.2 (3.4)

6. Secondary Outcome: Change From Baseline in FPG (Week 68)
Description: Change from baseline (week 0) in FPG was evaluated at week 68. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of additional anti-diabetic medication or discontinuation of trial treatment.
Time Frame: Baseline (week 0), week 68
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Oral Semaglutide 14 mg | Oral Semaglutide 25 mg | Oral Semaglutide 50 mg
Number analyzed (Participants) | 485 | 466 | 485
mmol/L | -2.4 (3.4) | -3.0 (3.7) | -3.2 (3.4)

7. Secondary Outcome: Percentage of Participants Who Achieved HbA1c Less Than (<) 7.0 (Percent [%]) (Week 52)
Description: Percentage of participants who achieved HbA1c <7.0 % at week 52 are presented. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of additional anti-diabetic medication or discontinuation of trial treatment.
Time Frame: At week 52
Population: FAS which comprised all randomised participants.
Measure: Number; unit: Percentage of Participants
Arm/Group | Oral Semaglutide 14 mg | Oral Semaglutide 25 mg | Oral Semaglutide 50 mg
Number analyzed (Participants) | 536 | 535 | 535
Percentage of Participants | 39 | 50.5 | 63

8. Secondary Outcome: Percentage of Participants Who Achieved HbA1c < 7.0 % (Week 68)
Description: Percentage of participants who achieved HbA1c <7.0 % at week 68 are presented. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of additional anti-diabetic medication or discontinuation of trial treatment.
Time Frame: At week 68
Population: FAS which comprised all randomised participants.
Measure: Number; unit: Percentage of Participants
Arm/Group | Oral Semaglutide 14 mg | Oral Semaglutide 25 mg | Oral Semaglutide 50 mg
Number analyzed (Participants) | 536 | 535 | 535
Percentage of Participants | 39.2 | 49.9 | 58.9

9. Secondary Outcome: Percentage of Participants Who Achieved HbA1c Less Than or Equal to (<=) 6.5 % (Week 52)
Description: Percentage of participants who achieved HbA1c <=6.5 % at week 52 are presented. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of additional anti-diabetic medication or discontinuation of trial treatment.
Time Frame: At week 52
Population: FAS which comprised all randomised participants.
Measure: Number; unit: Percentage of Participants
Arm/Group | Oral Semaglutide 14 mg | Oral Semaglutide 25 mg | Oral Semaglutide 50 mg
Number analyzed (Participants) | 536 | 535 | 535
Percentage of Participants | 25.8 | 39.6 | 51.2

10. Secondary Outcome: Percentage of Participants Who Achieved HbA1c <= 6.5 % (Week 68)
Description: Percentage of participants who achieved HbA1c <=6.5 % at week 68 are presented. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of additional anti-diabetic medication or discontinuation of trial treatment.
Time Frame: At week 68
Population: FAS which comprised all randomised participants.
Measure: Number; unit: Percentage of Participants
Arm/Group | Oral Semaglutide 14 mg | Oral Semaglutide 25 mg | Oral Semaglutide 50 mg
Number analyzed (Participants) | 536 | 535 | 535
Percentage of Participants | 23.6 | 35.8 | 46.2

11. Secondary Outcome: Time to Event Analyses of Rescue Medication
Description: Time to event analyses of rescue medication was evaluated from baseline (week 0) to week 68. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of additional anti-diabetic medication or discontinuation of trial treatment.
Time Frame: Baseline (week 0), week 68
Population: as for outcome 2
Measure: Median (Full Range); unit: Weeks
Arm/Group | Oral Semaglutide 14 mg | Oral Semaglutide 25 mg | Oral Semaglutide 50 mg
Number analyzed (Participants) | 92 | 54 | 48
Weeks | NA [NA to NA] — Due to insufficient number of participants with events to calculate via Kaplan Meir, data was not estimable. | NA [NA to NA] — Due to insufficient number of participants with events to calculate via Kaplan Meir, data was not estimable. | NA [NA to NA] — Due to insufficient number of participants with events to calculate via Kaplan Meir, data was not estimable.

12. Secondary Outcome: Change From Baseline in Body Weight (Week 68)
Description: Change from baseline (week 0) in body weight was evaluated at week 68. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of additional anti-diabetic medication or discontinuation of trial treatment.
Time Frame: Baseline (week 0), week 68
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Oral Semaglutide 14 mg | Oral Semaglutide 25 mg | Oral Semaglutide 50 mg
Number analyzed (Participants) | 495 | 477 | 495
Kg | -4.5 (5.5) | -7.1 (7.4) | -8.2 (8.1)

13. Secondary Outcome: Percentage Change From Baseline in Body Weight (Week 52)
Description: Percentage change from baseline (week 0) in body weight was evaluated at week 52. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of additional anti-diabetic medication or discontinuation of trial treatment.
Time Frame: Baseline (week 0), week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage change in body weight
Arm/Group | Oral Semaglutide 14 mg | Oral Semaglutide 25 mg | Oral Semaglutide 50 mg
Number analyzed (Participants) | 503 | 480 | 495
Percentage change in body weight | -4.7 (5.4) | -7.3 (6.6) | -8.5 (7.3)

14. Secondary Outcome: Percentage Change From Baseline in Body Weight (Week 68)
Description: Percentage change from baseline (week 0) in body weight was evaluated at week 68. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of additional anti-diabetic medication or discontinuation of trial treatment.
Time Frame: Baseline (week 0), week 68
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage change in body weight
Arm/Group | Oral Semaglutide 14 mg | Oral Semaglutide 25 mg | Oral Semaglutide 50 mg
Number analyzed (Participants) | 495 | 477 | 495
Percentage change in body weight | -4.7 (5.6) | -7.2 (7.1) | -8.4 (7.7)

15. Secondary Outcome: Percentage Change From Week 12 in Body Weight (Week 52)
Description: Percentage change in body weight was evaluated from week 12 to week 52. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of additional anti-diabetic medication or discontinuation of trial treatment.
Time Frame: Week 12, Week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage change in body weight
Arm/Group | Oral Semaglutide 14 mg | Oral Semaglutide 25 mg | Oral Semaglutide 50 mg
Number analyzed (Participants) | 370 | 366 | 355
Percentage change in body weight | -1.5 (3.6) | -3.8 (5.4) | -5.4 (6.1)

16. Secondary Outcome: Change From Baseline in Body Mass Index (BMI) (Week 52)
Description: Change from baseline (week 0) in body mass index (BMI) was evaluated at week 52. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of additional anti-diabetic medication or discontinuation of trial treatment.
Time Frame: Baseline (week 0), week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kilogram per square metre (kg/m^2)
Arm/Group | Oral Semaglutide 14 mg | Oral Semaglutide 25 mg | Oral Semaglutide 50 mg
Number analyzed (Participants) | 503 | 480 | 495
kilogram per square metre (kg/m^2) | -1.6 (1.8) | -2.5 (2.5) | -2.9 (2.6)

17. Secondary Outcome: Change From Baseline in BMI (Week 68)
Description: Change from baseline (week 0) in BMI was evaluated at week 68. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of additional anti-diabetic medication or discontinuation of trial treatment.
Time Frame: Baseline (week 0), week 68
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Oral Semaglutide 14 mg | Oral Semaglutide 25 mg | Oral Semaglutide 50 mg
Number analyzed (Participants) | 495 | 477 | 495
kg/m^2 | -1.6 (1.9) | -2.5 (2.7) | -2.9 (2.8)

18. Secondary Outcome: Change From Baseline in Waist Circumference (Week 52)
Description: Change from baseline (week 0) in waist circumference was evaluated at week 52. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of additional anti-diabetic medication or discontinuation of trial treatment.
Time Frame: Baseline (week 0), week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: centimetre (cm)
Arm/Group | Oral Semaglutide 14 mg | Oral Semaglutide 25 mg | Oral Semaglutide 50 mg
Number analyzed (Participants) | 502 | 479 | 494
centimetre (cm) | -4 (7) | -5 (7) | -6 (7)

19. Secondary Outcome: Change From Baseline in Waist Circumference (Week 68)
Description: Change from baseline (week 0) in waist circumference was evaluated at week 68. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of additional anti-diabetic medication or discontinuation of trial treatment.
Time Frame: Baseline (week 0), week 68
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Oral Semaglutide 14 mg | Oral Semaglutide 25 mg | Oral Semaglutide 50 mg
Number analyzed (Participants) | 494 | 476 | 495
cm | -4 (6) | -6 (7) | -7 (8)

20. Secondary Outcome: Percentage of Participants Who Achieved Weight Loss Greater Than or Equal to (>=) 5 % (Week 52)
Description: Percentage of participants who achieved weight loss >= 5 % at week 52 are presented. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of additional anti-diabetic medication or discontinuation of trial treatment.
Time Frame: At week 52
Population: FAS which comprised all randomised participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Oral Semaglutide 14 mg | Oral Semaglutide 25 mg | Oral Semaglutide 50 mg
Number analyzed (Participants) | 536 | 535 | 535
Percentage of participants | 41 | 60 | 67.5

21. Secondary Outcome: Percentage of Participants Who Achieved Weight Loss >= 5 % (Week 68)
Description: Percentage of participants who achieved weight loss >= 5 % at week 68 are presented. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of additional anti-diabetic medication or discontinuation of trial treatment.
Time Frame: At week 68
Population: FAS which comprised all randomised participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Oral Semaglutide 14 mg | Oral Semaglutide 25 mg | Oral Semaglutide 50 mg
Number analyzed (Participants) | 536 | 535 | 535
Percentage of participants | 42.2 | 58.5 | 65.7

22. Secondary Outcome: Percentage of Participants Who Achieved Weight Loss >= 10 % (Week 52)
Description: Percentage of participants who achieved weight loss >= 10 % at week 52 are presented. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of additional anti-diabetic medication or discontinuation of trial treatment.
Time Frame: At week 52
Population: FAS which comprised all randomised participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Oral Semaglutide 14 mg | Oral Semaglutide 25 mg | Oral Semaglutide 50 mg
Number analyzed (Participants) | 536 | 535 | 535
Percentage of participants | 13.9 | 29 | 37.2

23. Secondary Outcome: Percentage of Participants Who Achieved Weight Loss >= 10 % (Week 68)
Description: Percentage of participants who achieved weight loss >= 10 % at week 68 are presented. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of additional anti-diabetic medication or discontinuation of trial treatment.
Time Frame: At week 68
Population: FAS which comprised all randomised participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Oral Semaglutide 14 mg | Oral Semaglutide 25 mg | Oral Semaglutide 50 mg
Number analyzed (Participants) | 536 | 535 | 535
Percentage of participants | 14.3 | 29.4 | 34.7

24. Secondary Outcome: Change From Baseline in Total Cholesterol (Week 52)
Description: Change from baseline (week 0) in total cholesterol was evaluated at week 52. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of additional anti-diabetic medication or discontinuation of trial treatment.
Time Frame: Baseline, Week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Oral Semaglutide 14 mg | Oral Semaglutide 25 mg | Oral Semaglutide 50 mg
Number analyzed (Participants) | 490 | 467 | 486
mmol/L | -0.04 (0.96) | -0.15 (1.10) | -0.06 (0.94)

25. Secondary Outcome: Change From Baseline in Total Cholesterol (Week 68)
Description: Change from baseline (week 0) in total cholesterol was evaluated at week 68. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of additional anti-diabetic medication or discontinuation of trial treatment.
Time Frame: Baseline, Week 68
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Oral Semaglutide 14 mg | Oral Semaglutide 25 mg | Oral Semaglutide 50 mg
Number analyzed (Participants) | 484 | 470 | 487
mmol/L | -0.03 (0.99) | -0.08 (1.05) | -0.06 (1.00)

26. Secondary Outcome: Change From Baseline in Low Density Lipoproteins (LDL) (Week 52)
Description: Change from baseline (week 0) in LDL was evaluated at week 52. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of additional anti-diabetic medication or discontinuation of trial treatment.
Time Frame: Baseline, Week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Oral Semaglutide 14 mg | Oral Semaglutide 25 mg | Oral Semaglutide 50 mg
Number analyzed (Participants) | 477 | 454 | 473
mmol/L | 0.04 (0.75) | -0.01 (0.85) | 0.11 (0.76)

27. Secondary Outcome: Change From Baseline in LDL (Week 68)
Description: Change from baseline (week 0) in LDL was evaluated at week 68. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of additional anti-diabetic medication or discontinuation of trial treatment.
Time Frame: Baseline, Week 68
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Oral Semaglutide 14 mg | Oral Semaglutide 25 mg | Oral Semaglutide 50 mg
Number analyzed (Participants) | 472 | 459 | 476
mmol/L | 0.07 (0.80) | 0.06 (0.85) | 0.08 (0.79)

28. Secondary Outcome: Change From Baseline in High Density Lipoproteins (HDL) (Week 52)
Description: Change from baseline (week 0) in HDL was evaluated at week 52. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of additional anti-diabetic medication or discontinuation of trial treatment.
Time Frame: Baseline, Week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Oral Semaglutide 14 mg | Oral Semaglutide 25 mg | Oral Semaglutide 50 mg
Number analyzed (Participants) | 477 | 453 | 474
mmol/L | 0.06 (0.18) | 0.07 (0.19) | 0.08 (0.18)

29. Secondary Outcome: Change From Baseline in HDL (Week 68)
Description: Change from baseline (week 0) in HDL was evaluated at week 68. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of additional anti-diabetic medication or discontinuation of trial treatment.
Time Frame: Baseline, Week 68
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Oral Semaglutide 14 mg | Oral Semaglutide 25 mg | Oral Semaglutide 50 mg
Number analyzed (Participants) | 473 | 458 | 476
mmol/L | 0.06 (0.19) | 0.08 (0.21) | 0.09 (0.20)

30. Secondary Outcome: Change From Baseline in Triglycerides (Week 52)
Description: Change from baseline (week 0) in triglycerides was evaluated at week 52. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of additional anti-diabetic medication or discontinuation of trial treatment.
Time Frame: Baseline, Week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Oral Semaglutide 14 mg | Oral Semaglutide 25 mg | Oral Semaglutide 50 mg
Number analyzed (Participants) | 489 | 465 | 483
mmol/L | -0.46 (1.77) | -0.65 (2.08) | -0.71 (1.40)

31. Secondary Outcome: Change From Baseline in Triglycerides (Week 68)
Description: Change from baseline (week 0) in triglycerides was evaluated at week 68. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of additional anti-diabetic medication or discontinuation of trial treatment.
Time Frame: Baseline, Week 68
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Oral Semaglutide 14 mg | Oral Semaglutide 25 mg | Oral Semaglutide 50 mg
Number analyzed (Participants) | 483 | 469 | 486
mmol/L | -0.51 (1.77) | -0.65 (2.06) | -0.70 (1.43)

32. Secondary Outcome: Number of Adverse Events
Description: An adverse event (AE) defined as any unfavourable and unintended sign, including an abnormal laboratory finding, symptom or disease (new or exacerbated) temporally associated with the use of an investigational medicinal products (IMP). Results are based on the data from the on-treatment observation period, which was the time period when a participant was on trial treatment, including any period after initiation of rescue medication.
Time Frame: From baseline (week 0) up to week 73
Population: Safety Analysis Set (SAS) which comprised all participants who received at least 1 dose of trial treatment. Overall number of participants analyzed = participants with available data for this outcome measure.
Measure: Number; unit: Events
Arm/Group | Oral Semaglutide 14 mg | Oral Semaglutide 25 mg | Oral Semaglutide 50 mg
Number analyzed (Participants) | 534 | 534 | 534
Events | 1641 | 2055 | 2115

33. Secondary Outcome: Number of Clinically Significant Hypoglycaemic Episodes (Level 2) (<3.0 mmol/L (54 Milligram Per Decilitre [mg/dL]) or Severe Hypoglycaemic Episodes (Level 3)
Description: Hypoglycaemic episodes were classified according to the American Diabetes Association 2018/ International Hypoglycaemia Study Group 2017, where glycemic criteria for level 2 was < 3.0 mmol/L (54 mg/dL) and level 3 had no specific glucose threshold. Results are based on the data from the on-treatment observation period, which was the time period when a participant was on trial treatment, including any period after initiation of rescue medication.
Time Frame: From baseline (week 0) up to week 68
Population: SAS which comprised all participants who received at least 1 dose of trial treatment. Overall number of participants analyzed = participants with available data for this outcome measure.
Measure: Number; unit: Count of episodes
Arm/Group | Oral Semaglutide 14 mg | Oral Semaglutide 25 mg | Oral Semaglutide 50 mg
Number analyzed (Participants) | 534 | 534 | 534
Count of episodes
  Level 2 | 65 | 44 | 35
  Level 3 | 0 | 0 | 1

34. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (Week 52)
Description: Change from baseline (week 0) in systolic blood pressure at week 52 are presented. Results are based on the data from the on-treatment observation period, which was the time period when a participant was on trial treatment, including any period after initiation of rescue medication.
Time Frame: Baseline (week 0), week 52
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: millimetres of mercury (mmHg)
Arm/Group | Oral Semaglutide 14 mg | Oral Semaglutide 25 mg | Oral Semaglutide 50 mg
Number analyzed (Participants) | 456 | 426 | 434
millimetres of mercury (mmHg) | -4 (14) | -6 (13) | -6 (14)

35. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (Week 68)
Description: Change from baseline (week 0) in systolic blood pressure at week 68 are presented. Results are based on the data from the on-treatment observation period, which was the time period when a participant was on trial treatment, including any period after initiation of rescue medication.
Time Frame: Baseline (week 0), week 68
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Oral Semaglutide 14 mg | Oral Semaglutide 25 mg | Oral Semaglutide 50 mg
Number analyzed (Participants) | 442 | 414 | 429
mmHg | -4 (13) | -6 (13) | -5 (13)

36. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure (Week 52)
Description: Change from baseline (week 0) in diastolic blood pressure at week 52 are presented. Results are based on the data from the on-treatment observation period, which was the time period when a participant was on trial treatment, including any period after initiation of rescue medication.
Time Frame: Baseline (week 0), week 52
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Oral Semaglutide 14 mg | Oral Semaglutide 25 mg | Oral Semaglutide 50 mg
Number analyzed (Participants) | 456 | 426 | 434
mmHg | -2 (8) | -2 (8) | -2 (8)

37. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure (Week 68)
Description: Change from baseline (week 0) in diastolic blood pressure at week 68 are presented. Results are based on the data from the on-treatment observation period, which was the time period when a participant was on trial treatment, including any period after initiation of rescue medication.
Time Frame: Baseline (week 0), week 68
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Oral Semaglutide 14 mg | Oral Semaglutide 25 mg | Oral Semaglutide 50 mg
Number analyzed (Participants) | 442 | 414 | 429
mmHg | -3 (8) | -3 (8) | -2 (8)

38. Secondary Outcome: Change From Baseline in Pulse (Week 52)
Description: Change from baseline (week 0) in pulse at week 52 are presented. Results are based on the data from the on-treatment observation period, which was the time period when a participant was on trial treatment, including any period after initiation of rescue medication.
Time Frame: Baseline (week 0), week 52
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: beats per minute (beats/min)
Arm/Group | Oral Semaglutide 14 mg | Oral Semaglutide 25 mg | Oral Semaglutide 50 mg
Number analyzed (Participants) | 456 | 426 | 434
beats per minute (beats/min) | 2 (10) | 2 (10) | 3 (11)

39. Secondary Outcome: Change From Baseline in Pulse (Week 68)
Description: Change from baseline (week 0) in pulse at week 68 are presented. Results are based on the data from the on-treatment observation period, which was the time period when a participant was on trial treatment, including any period after initiation of rescue medication.
Time Frame: Baseline (week 0), week 68
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Oral Semaglutide 14 mg | Oral Semaglutide 25 mg | Oral Semaglutide 50 mg
Number analyzed (Participants) | 442 | 413 | 429
beats/min | 1 (10) | 2 (10) | 2 (10)

ADVERSE EVENTS:
Time Frame: Week 0 to week 73
Description: Serious adverse events and other AEs were based on the on-treatment observation period, i.e., time period when a participant was on treatment with trial product, including any period after initiation of rescue medication. All-cause mortality were based on the in-trial observation period, i.e., the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of additional anti-diabetic medication or discontinuation of trial treatment.
Arm/Group | Oral Semaglutide 14 mg | Oral Semaglutide 25 mg | Oral Semaglutide 50 mg
All-Cause Mortality (participants affected / at risk) | 2/534 | 6/534 | 2/534
Serious Adverse Events (participants affected / at risk) | 53/534 | 57/534 | 44/534
Other Adverse Events (participants affected / at risk) | 277/534 | 294/534 | 314/534
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Semaglutide 14 mg (N=534) | Oral Semaglutide 25 mg (N=534) | Oral Semaglutide 50 mg (N=534)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abscess intestinal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Abscess oral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Acute left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 4 (4) | 3 (3) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Aortic valve disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Appendicitis perforated (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 1 (1) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Brachial plexus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 3 (3) | 0 (0) | 3 (3)
COVID-19 pneumonia (Infections and infestations) | 2 (2) | 2 (2) | 2 (2)
Calculus bladder (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Carotid artery occlusion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cataract subcapsular (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis pharyngeal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Central nervous system lesion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 1 (2) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Chronic coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Chronic myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Circulatory collapse (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Conduction disorder (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 2 (2) | 1 (1) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cystocele (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Diabetic gangrene (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Enterocele (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Epididymitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Epiretinal membrane (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 1 (3) | 0 (0) | 1 (1)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gallbladder disorder (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Glomerular filtration rate decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Greater trochanteric pain syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Gynaecomastia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Hip arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Iliac artery stenosis (Vascular disorders) | 0 (0) | 1 (2) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ischaemic skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Keratoplasty (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Macular oedema (Eye disorders) | 1 (2) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Myelopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Papilloedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal hypertension (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Somatic symptom disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Speech disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Splenic injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Swelling face (General disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Semaglutide 14 mg (N=534) | Oral Semaglutide 25 mg (N=534) | Oral Semaglutide 50 mg (N=534)
Abdominal pain (Gastrointestinal disorders) | 14 (25) | 27 (34) | 21 (27)
Abdominal pain upper (Gastrointestinal disorders) | 14 (17) | 32 (52) | 22 (55)
COVID-19 (Infections and infestations) | 63 (65) | 64 (68) | 66 (68)
Constipation (Gastrointestinal disorders) | 40 (46) | 35 (41) | 33 (39)
Decreased appetite (Metabolism and nutrition disorders) | 38 (43) | 39 (42) | 58 (61)
Diabetic retinopathy (Eye disorders) | 41 (44) | 26 (30) | 35 (40)
Diarrhoea (Gastrointestinal disorders) | 66 (84) | 69 (108) | 76 (150)
Dyspepsia (Gastrointestinal disorders) | 28 (32) | 29 (47) | 30 (50)
Headache (Nervous system disorders) | 34 (63) | 28 (81) | 38 (81)
Nasopharyngitis (Infections and infestations) | 24 (28) | 22 (27) | 27 (30)
Nausea (Gastrointestinal disorders) | 96 (119) | 145 (222) | 146 (218)
Vomiting (Gastrointestinal disorders) | 52 (69) | 91 (155) | 97 (184)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2022-09-16): https://cdn.clinicaltrials.gov/large-docs/69/NCT04707469/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-23): https://cdn.clinicaltrials.gov/large-docs/69/NCT04707469/SAP_001.pdf